CLINICAL TRIAL: NCT07146477
Title: From Markets to Meals: A Mixed Methods Study on How Urban Slum Food Environments Influence Caregivers' Feeding Practices for Children Under Five Years in Pune, India
Brief Title: A Mixed Methods Study on How Urban Slum Food Environments Influence Caregivers' Feeding Practices for Children Under Five Years in Pune, India
Acronym: FEFC
Status: Not yet recruiting | Type: Observational
Sponsor: Hirabai Cowasji Jehangir Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Anuradha Khadilkar, Deputy Director, Hirabai Cowasji Jehangir Medical Research Institute
Other Study IDs: MCH-FEFC-2025-07
Record Dates: First submitted 2025-08-16; First posted 2025-08-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Feeding Practices; Food Choices; Maternal and Child Health
Keywords: Food Choice Drivers; Food Environment; Urban Slums; India; Family; Infant Feeding

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Family or Household: Family or Households (n = 250) include all the members residing in one house sharing food and other amenities and who have children under 5 years of age.
- Food Vendors: Food Vendors (n = 120) who operate in the 500 m radius of the household cluster will be interviewed in depth to characterize the type of foods sold so that the food environment of the family can be characterized.

SUMMARY:
The goal of this observational study is to examine how urban slum food environments influence caregivers' feeding practices for children under five years of age in Pune. The main questions it aims to answer are:

* What are the characteristics of the food environment in selected slums of Pune using the 5 A's framework: availability, accessibility, affordability, acceptability, and accommodation?
* What are caregivers' perceptions of food safety, food prestige, and convenience as additional drivers of food choice within the slum context?
* Are caregivers' aware, and have understanding about the use of packaged food labels, especially in relation to identifying foods for young children?
* How do the local food environment and food choice (FEFC) drivers interact to influence caregivers' feeding practices, with a particular focus on the consumption of unhealthy foods and sugar-sweetened beverages among children under five years of age? Participants will be interviewed using digital forms to assess their food environment and food choice drivers. Anthropometric measurements of all children under five years of age in the household will be taken.

DETAILED DESCRIPTION:
In India there is a high prevalence of poor complementary feeding practices. Around 1 in 2 caregivers introduced complementary foods to infants at 6-8 months, while 1 in 4 infants had the minimum dietary diversity, and 1 in 10 consumed the minimum acceptable diet. A worrisome trend being observed is the widespread consumption of ultra-processed foods (UPFs) among children across all socioeconomic groups in India. In informal settlements in Mumbai, nearly 60% children under 6 years were found to be consuming UPFs daily. Increased UPF consumption contributes significantly to the prevalence of double burden of malnutrition in India.

Pune is a rapidly growing mega-city in Maharashtra with a population of 9.4 million, which includes over 1.2 million slum-dwellers, including around 300,000 children under-five years of age. In 2020, only 6% infants had adequate diets and 12% achieved dietary diversity. Specific data is lacking on time of introduction of complementary foods and no data are available on slum-dwelling populations. The United Nations Human Settlements Program defines a slum as "a group of individuals who live under the same roof, and that lack one or more of the following conditions: access to improved water, access to improved sanitation, sufficient living space, the durability of housing, and secure tenure". Slums are a unique and complex ecosystem where caregivers face multiple, intersecting challenges when making food choices for their children. These settings are often marked by limited infrastructure, economic constraints, and a high density of informal food vendors-conditions that may promote the availability and consumption of unhealthy foods.

The food environment defined as "consumer interface within the food system that encompasses the availability, affordability, convenience, quality and promotion, and sustainability of foods and beverages in wild, cultivated, and built spaces" is increasingly recognized as a key determinant of dietary behavior. Yet there is limited evidence from Indian slum settings on how food environments influence infant and young child feeding (IYCF) practices. Most existing research focuses on maternal knowledge or household-level factors, with minimal attention to the broader environmental and structural influences.

This study responds to this gap by assessing the 5 A's of the food environment (availability, accessibility, affordability, acceptability, and accommodation), and by exploring how these dimensions interact with caregivers' perceptions of convenience, food safety, and prestige, as well as their ability to understand and use food labels. These factors are particularly relevant in urban slums, where informal food systems dominate, and where unhealthy foods may be more readily available and aspirationally consumed. Therefore, the objectives of this study are:

1. To characterize the food environment in selected slums of Pune using the 5 A's framework: availability, accessibility, affordability, acceptability, and accommodation.
2. To explore caregivers' perceptions of food safety, food prestige, and convenience as additional drivers of food choice within the slum context.
3. To assess caregivers' awareness, understanding, and use of packaged food labels, especially in relation to identifying foods for young children.
4. To examine how the local food environment and food choice drivers interact to influence caregivers' feeding practices, with a particular focus on the consumption of unhealthy foods and sugar-sweetened beverages among children under five.
5. To disseminate findings through awareness sessions and cooking competitions.

ELIGIBILITY:
Inclusion Criteria:

* For Family Units:

  1. Families who had participated in the previous house-to-house survey to determine maternal healthcare utilization and infant and young child feeding practices.
  2. Families where all the female caregivers are willing to participate.
* For Food Vendors:

  1. Food vendors who regularly carry out business in the 500 m radius of the household.
  2. Willingness to participate in the study.

Exclusion Criteria:

* 1. Families who were a part of the earlier project but have moved out of the survey area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. The study population will consist of Infant and young child caregivers living in slums who have a child or children less than five years of age and had enrolled in an earlier study to assess utilization of maternal healthcare services in these slums.
  2. Food vendors (stores, mobile informal vendors and hawkers, and restaurants) who function in the 500 m radius of the household.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2025-09-29 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage food items in each of the 28 food groups available in each of the 4 study locations | An average of 1 year
  Food Availability in each study location will be assessed as the percentage food items available for purchase in each of the 28 food groups. The Food Outlet Census (https://sites.rutgers.edu/food-environment-toolbox/community-food-environment-mapping-food-outlet-census/) tool is being used to collect data on the foods available but the tool does not have any specific scoring criteria.
Percentage of families in each study location who can afford to buy a healthy diet | An average of 1 Year
  Food Affordability of families will be assessed as the percentage of families who can afford a healthy diet. For this purpose then investigators will calculate Cost of a Healthy Diet (CoHD) using the tool available from Tufts University: https://sites.tufts.edu/foodpricesfornutrition/tools/. Per capita income of each household will also be calculated. These two parameters will help the investigators calculate the percentage of families in each location who can afford a healthy diet.
Percentage of food items considered convenient by households in each location | An average of 1 year
  Convenience will be assessed as percentage of food items in each of the 28 food groups which participants consider convenient because their ease of storage, low perishability, ease of preparation.
Gender and Family Role of the primary food-related decision maker | An average of 1 year
  The gender and family role of primary food-related decision maker will be assessed as percentages and illustrated using pie-charts
Percentage of participants concerned with food safety | An average of 1 year
  Percentage of participants worried of safety of food due to poor hygiene or use of pesticides will be asessed
Percentage of households with label awareness | An average of 1 year
  The percentage of households who were aware of food labeling (read labels, knew where the label was located) will be assessed
Correlation of food environment characteristics with infant and young child feeding practices | An average of 1 year
  The correlation of different food environment characteristics such as accessibility, availability, affordability, with infant and young child feeding indicators such as ultra-processed food consumption, zero fruit and vegetable consumption

SECONDARY OUTCOMES:
Number and types of food outlets in the study location | An average of 1 year
  The number and types (grocery, wholesaler, specialty stores, etc) in the study location will be calculated and presented.
Type of foods being promoted in the study locations | An average of 1 year
  The type of foods being promoted by roadside promotions in the study locations will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hirabai Cowasji Jehangir Medical Research Institute, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
Pseudonymized individual participant data (IPD) will be shared upon reasonable request made to the Principal Investigator only after primary study publications have been completed.